CLINICAL TRIAL: NCT07196384
Title: Optical PD-1 and PD-L1 Imaging Using Dual-wavelength Quantitative Fluorescence Endoscopy in Locally Advanced Esophageal Cancer Using Durvalumab-680LT and Nivolumab-800CW
Brief Title: Optical PD-1 and PD-L1 Imaging in Locally Advanced Esophageal Cancer Using Durvalumab-680LT and Nivolumab-800CW
Acronym: GLOW
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Martini Hospital Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMCG 21164; 2024-520090-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-22; First posted 2025-09-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 mg durvalumab-680LT + 15 mg nivolumab-800CW in esophageal cancer (Experimental)
  Interventions: Device: Spectroscopy system; Drug: Nivolumab-800CW; Drug: Durvalumab-680LT
- 25 mg durvalumab-680LT + 25 mg nivolumab-800CW in esophageal cancer (Experimental)
  Interventions: Device: Spectroscopy system; Drug: Nivolumab-800CW; Drug: Durvalumab-680LT

INTERVENTIONS:
Device: Spectroscopy system — System that measures the fluorescence intensity in tissue in vivo.
Drug: Nivolumab-800CW — Fluorescent tracer
Drug: Durvalumab-680LT — Fluorescent tracer

SUMMARY:
Radiation and chemotherapy can shrink the tumor. For certain types of cancer, immunotherapy is added to further reduce the tumor size. Immunotherapy works for some patients and can sometimes keep the cancer under control for a long time. Unfortunately, immunotherapy does not work for every patient. That's why researchers around the world are looking for new ways to predict who will benefit from immunotherapy and who will not.

It is likely that immunotherapy is more effective when the tumor or immune cells have specific targets, such as the proteins PD-L1 or PD-1. Unfortunately, clinicians cannot reliably detect these proteins through blood tests or tissue samples, because their presence can vary throughout the tumor.

With this study, the investigators hope to use a new technique called 'fluorescence endoscopy' during an endoscopic ultrasound of the esophagus to visualize whether the PD-L1 or PD-1 proteins are present in esophageal cancer or immune cells. Additionally, the investigators aim to investigate whether the presence of these proteins changes before and after chemotherapy and/or radiation. This will help us determine the best timing for measuring these proteins in the future.

What is fluorescence endoscopy? To determine whether the proteins are present, participants in this study will receive two 'tracers' via an IV beforehand. The first tracer is a fluorescent substance-a kind of 'glow-in-the-dark' compound-attached to a drug that binds to PD-L1 proteins in esophageal cancer. The second fluorescent tracer binds to PD-1 proteins on immune cells.

During fluorescence endoscopy, the investigators use special equipment to detect these tracers in the esophagus. This information may help us better identify which patients are suitable for immunotherapy treatment and which are not.

ELIGIBILITY:
Inclusion Criteria:

* Lesion suspected for locally advanced EC (cT1b-4a N0-3 M0);
* Indication for neoadjuvant therapy or definitive chemo-radiation therapy;
* Age ≥ 18 years;
* Written informed consent.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent according to treating medical physician;
* Concurrent uncontrolled medical conditions according to treating medical physician;
* Medical history of auto-immune disease and on active treatment;
* Pregnancy or breast feeding. A negative pregnancy test must be available for women of childbearing potential (i.e. premenopausal women with intact reproductive organs and women less than two years after menopause);
* Irradical endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) of the primary tumor prior to start of neoadjuvant therapy according to the patient's medical history;
* Received an investigational drug within 30 days prior to the tracer administration according to the patient's medical history;
* History of infusion reactions to durvalumab or nivolumab or other monoclonal antibodies according to the patient's medical history;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasiblity | Up to 14 months
  To determine the feasibility of our newly built dual-wavelength spectroscopy system in combination with the fluorescent tracers durvalumab-680LT and nivolumab-800CW. The spectroscopy system is considered feasible if at least 4 out of 10 patients demonstrate a higher tumor-to-healthy tissue ratio based on spectroscopy measurements. This ratio is calculated by dividing the spectroscopy value of the tumor region by that of the adjacent healthy tissue. The threshold of 4 out of 10 patients was selected based on literature data, which indicate that approximately 43.5% to 48.1% of patients exhibit high PD-1/PD-L1 expression in the tumor area. The investigators therefore expect a similar proportion of patients to show elevated spectroscopy values corresponding to increased target expression.
Safety of dual tracer administratio | Up to 14 months
  • To assess the safety of dual tracer administration of nivolumab-800CW and durvalumab-680LT by evaluating heart rate in beats per minute.

SECONDARY OUTCOMES:
Safety of dual tracer administration | Up to 14 months
  • To assess the safety of dual tracer administration of nivolumab-800CW and durvalumab-680LT by evaluating blood pressure in mmHg
Safety of dual tracer administration | Up to 14 months
  To assess the safety of dual tracer administration of nivolumab-800CW and durvalumab-680LT by evaluating number of AE's
Safety of dual tracer administration | Up to 14 months
  To assess the safety of dual tracer administration of nivolumab-800CW and durvalumab-680LT by evaluating number of SAE'S
Safety of dual tracer administration | Up to 14 months
  To assess the safety of dual tracer administration of nivolumab-800CW and durvalumab-680LT by evaluating number of SUSARS.
Correlation between in vivo signal and ex vivo pathology | Up to 14 months
  • To investigate the correlation between fluorescence signals detected in vivo with ex vivo histopathology, immunohistochemistry; This correlation will be measured by comparing the percentage of staining on immunohistochemistry staining and the hight of the fluorescence signals detected in vivo (unit: Q • μfa,x).
Correlation of fluorescence intensity before and after neoadjuvant therapy | Up to 14 months
  • To compare the fluorescence intensity of the fluorescent tracer durvalumab-680LT and nivolumab-800CW before and after neoadjuvant therapy. These measurements will be taken with a spectroscopy device at two different time points. The first before neoadjuvant treatment, the second after neoadjuvant treatment. The unit of the fluorescence intensity is Q • μfa,x. Both measurements will be compared with each other.
Correlation between in vivo signal and ex vivo analysis | Up to 14 months
  • To compare fluorescence signals detected in vivo taken with a spectroscopy device during study-specific procedures with the percentage of fluorescence staining assessed by fluorescence microscopy
Investigate the sub-cellular location of the drugs. | Up to 14 months
  • To assess the (sub)-cellular location and distribution of durvalumab-680LT and nivolumab-800CW by ex vivo fluorescence microscopy. The investigators image a slide of a biopsy block with the fluorescence microscope, after imaging the investigators introduce fluorescence markers targeting certain cell types on the same slide. These slides can be imaged with the fluorescence microscope again. Afterwards the two slides can be compared with each other to look for overlap.
Optimal dose determination of nivolumab-800CW | up to 12 months
  • To determine the most optimal dose of nivolumab-800CW for fluorescence molecular endoscopy.

IPD SHARING:
Plan to Share IPD: No